CLINICAL TRIAL: NCT07299019
Title: A Phase 3, Randomized, Double-blind, Efficacy and Safety Study Comparing Orelabrutinib to Placebo in Patients With Non-active Secondary Progressive Multiple Sclerosis
Brief Title: A Study of Orelabrutinib in Patients With Secondary Progressive Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB020-03-002
Record Dates: First submitted 2025-12-18; First posted 2025-12-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib Group (Experimental): Orelabrutinib PO daily
  Interventions: Drug: Orelabrutinib
- Placebo Group (Placebo Comparator): Placebo PO daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib orally
  Arms: Orelabrutinib Group
Drug: Placebo — Placebo orally
  Arms: Placebo Group

SUMMARY:
Orelabrutinib is a CNS-penetrable BTK inhibitor. This is a phase 3, randomized, double-blind, parallel-group, multicenter study to evaluate the efficacy and safety of orelabrutinib compared with placebo in patients with non-active Secondary Progress MS. Patients will be treated for approximately 24 to 60 months, with a minimum treatment duration of 12 months. The study will enroll approximately 990 subjects in a 2:1 randomization (orelabrutinib: placebo), globally.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, parallel-group, multicenter study to evaluate the efficacy and safety of orelabrutinib compared with placebo in patients with naSPMS. The study will enroll approximately 990 subjects in a 2:1 randomization (orelabrutinib: placebo), globally.

The study consists of the following periods:

* Screening Period: Up to 4 weeks.
* Treatment Period: The duration of treatment will vary for individual participants ranging from approximately 24 to 60 months, depending on the time of recruitment. A month is defined as a period of 28 days by convention.
* Double-blinded (DB) Treatment: All eligible participants will be randomized at 2:1 ratio to accept orelabrutinib QD or placebo during the DB treatment period. The study will be unblinded when all participants in the DB period have reached a minimum treatment duration of 12 months at the time of primary analysis timing cutoff.
* Open-label (OL) Treatment: Participants with 24-week CDP as assessed by EDSS are eligible for 2-year open-label orelabrutinib treatment.
* Safety Follow-Up Period: It will last 4 weeks. The safety follow-up period will begin when the participants discontinue from the treatment before the end of the trial for any reasons or complete the trial but do not enter the long-term safety study (LTS) (see below).

All active study participants will have a final end of study (EOS) visit within 4 weeks of the study end date. Participants who are receiving IMP in DB or OL but do not consent to or are not eligible for enrollment in the LTS study, must return for a final safety follow-up visit 4 weeks later. For participants who intend and are eligible to join the LTS, open-label treatment with orelabrutinib will continue and no safety follow-up will occur.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years of age, inclusive, at the time of signing the informed consent.
2. Participant must have a previous diagnosis of RRMS in accordance with 2024 McDonald criteria
3. Participant must have a current diagnosis of SPMS in accordance with the clinical course criteria revised in 2013
4. Participant must have documented evidence of disability progression independent of clinical relapse observed during the 24 months before screening. A written summary of the clinical evidence of disability progression must be discussed and aligned between the Investigator and the Sponsor's dedicated qualified person(s).
5. Absence of clinical relapses for at least 24 months.

Exclusion Criteria:

1. The patient has been diagnosed with primary progressive MS (PPMS) according to 2024 McDonald diagnostic criteria
2. Immunologic disorder other than MS or any other conditions requiring corticosteroid therapy.
3. History or current diagnosis of other neurological disorders that may mimic MS
4. History or current diagnosis of progressive multifocal leukoencephalopathy
5. Active, clinically significant viral, bacterial, or fungal infection
6. History of any other significant active medical condition
7. History of suicidal behavior within 6 months prior to Screening
8. Any prior history of malignancy
9. Patients on anticoagulation, or antiplatelet therapy
10. Patients took strong/moderate CYP3A inhibitors or strong/moderate CYP3A inducers within 14 days
11. Clinically significant laboratory abnormalities at Screening.
12. Vaccination with live or live-attenuated virus vaccine within 1 month prior to Screening
13. History of alcohol abuse or alcohol use disorder or other drug abuse within 12 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 990 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Time to onset of confirmed disability progression (CDP) events, confirmed over at least 24 weeks | Up to approximately 120 weeks
  Expanded disability status scale (EDSS) score increase ≥ 1.0 point from baseline when the baseline score is ≤ 5.0, or ≥ 0.5 points from baseline when the baseline score is > 5.0

SECONDARY OUTCOMES:
12 Week CDP | Up to approximately 120 weeks
  Time to onset of CDP events on EDSS, confirmed over at least 12 weeks
T2 lesions on MRI | Up to approximately 120 weeks
  The total number of new or enlarging T2 lesions on MRI scans of the brain
24-week CDP-9-hole Peg Test | Up to approximately 120 weeks
  Time to onset of CDP events on 9-hole Peg Test (9HPT), defined as ≥ 20% increase on 9HPT from baseline, confirmed over at least 24 weeks
24-week CDP-T25FWT | Up to approximately 120 weeks
  Time to onset of CDP events on Timed 25-Foot Walk Test (T25FWT), defined as ≥ 20% increase on T25FWT from baseline, confirmed over at least 24 weeks
24-week CDI | Up to approximately 120 weeks
  Time to onset of confirmed disability improvement (CDI) events on EDSS, defined as ≥ 1.0-point decrease on the EDSS score from baseline when the baseline score is ≤ 5.0, or ≥ 0.5 points from baseline when the baseline score is > 5.0, confirmed over at least 24 weeks
24-week CDI-9HPT | Up to approximately 120 weeks
  Time to onset of CDI events on 9HPT, defined as ≥ 20% decrease on the 9HPT score from baseline, confirmed over at least 24 weeks
24-week CDI-T25FWT | Up to approximately 120 weeks
  Time to onset of CDI events on T25FWT, defined as ≥ 20% decrease on the T25FWT score from baseline, confirmed over at least 24 weeks
Symbol Digit Modalities Test | Up to approximately 120 weeks
  The change in cognitive function as assessed by Symbol Digit Modalities Test (SDMT) from baseline to each scheduled visit
Annualized relapse rate | Up to approximately 120 weeks
  Annualized relapse rate (ARR) during the study period assessed by protocol-defined adjudicated relapses
To evaluate the safety and tolerability of orelabrutinib | Up to approximately 120 weeks
  Safety as assessed by the nature, severity, and incidence of adverse events (AEs) (graded according to National Cancer Institute-Common Terminology Criteria for AEs, NCI-CTCAE version 5.0);